CLINICAL TRIAL: NCT01240694
Title: An Open-Label Long-Term Study of the Safety and Tolerability of Repeated Administration of CEP-33457 in Patients With Systemic Lupus Erythematosus
Brief Title: A Long-Term Study of the Safety and Tolerability of Repeated Administration of CEP-33457 in Participants With Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision; there were no safety issues
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C33457/3075
Record Dates: First submitted 2010-10-15; First posted 2010-11-15 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — spliceosomal peptide P140

ARMS (1):
- CEP-33457 (Experimental): Participants will receive 200 micrograms (mcg) of CEP-33457
  Interventions: Drug: CEP-33457

INTERVENTIONS:
Drug: CEP-33457 — CEP-33457 will be administered subcutaneously per dose specified in the arm description.
  Other Names: Lupuzor

SUMMARY:
The primary objective of this study is to evaluate the long term safety and tolerability of repeated administration of subcutaneous (SC) CEP-33457 for injection every 4 weeks over 72 weeks (18 doses) in participants with systemic lupus erythematosus (SLE) who have participated in a previous Cephalon sponsored clinical study of CEP-33457, and completed at least Visit 8 (Week 24 of that study).

ELIGIBILITY:
Inclusion Criteria:

* The participant has an established diagnosis of SLE as defined by ACR Classification Revised Criteria. The diagnosis is fulfilled provided that at least 4 criteria are met.
* The participant previously participated in and completed at least Visit 8 (Week 24) the Cephalon sponsored clinical study with CEP-33457 (study C33457/2047) and, in the investigator's opinion, would benefit from continued participation in a clinical study.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of contraception, and must agree to continued use of this method for the duration of the study and for 30 days after discontinuation of study drug treatment.

Exclusion Criteria:

* The participant has New York Heart Association (NYHA) Class III or IV congestive heart failure.
* The participant has an estimated glomerular filtration rate (eGFR) of less than 30 milliliters (mL)/minute (min)/1.73 square meter (m^2) (via Modification of Diet in Renal Disease [MDRD] equation).
* The participant has an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value greater than 2 times the upper limit of normal (ULN) or a total bilirubin level greater than 1.5 times ULN.
* The participant has a planned immunization with a live or live attenuated vaccine within 3 months prior to administration of the first dose of study drug and for 3 months after administration of the last dose of study drug.
* The participant has any clinically significant abnormalities on electrocardiogram (ECG) that are not related to SLE, as determined by the investigator. Participants with stable ECG changes without evidence of active cardiovascular disease may participate at the discretion of the investigator and medical monitor.
* The participant has an ongoing active systemic infection requiring treatment or a history of severe infection, such as hepatitis or pneumonia, in the 3 months prior to administration of the first dose of study drug. Less severe infections in the 3 months prior to administration of the first dose of study drug are permitted at the discretion of the investigator and medical monitor.
* The participant has any concomitant medical condition unrelated to SLE that may interfere with his or her safety or with evaluation of the study drug, as determined by the investigator.
* The participant has a history of a positive test result for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab).
* The participant has a known positive history of antibodies to human immunodeficiency virus (HIV) or HIV disease.
* The participant has a history of alcohol or substance dependence or abuse (with the exception of nicotine), according to the Diagnostic and Statistical Manual of Mental Disorders of the American Psychiatric Association, Fourth Edition, Text Revision (DSM-IV-TR), within 3 months of the screening visit for study C33457/2047, or has current substance abuse.
* The participant has a history of severe allergic reactions to or hypersensitivity to any component of the study drug.
* The participant is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The participant has undergone or is undergoing treatment with another investigational drug for the treatment of lupus within 6 months prior to the 1st dose of study drug or has received any other investigational drug for any other condition within 30 days prior to the 1st dose of study drug, except for treatment with CEP-33457 or placebo in study C33457/2047.
* The participant has a known history of antibodies to CEP-33457.
* The participant is unlikely to comply with the study protocol or is unsuitable for any other reason, as judged by the investigator or medical monitor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-12-09 (Actual); Primary Completion 2012-06-14 (Actual); Study Completion 2012-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (85):
- United States (39):
  - Teva Investigational Site 27, Birmingham, Alabama
  - Teva Investigational Site 20, Tucson, Arizona
  - Teva Investigational Site 16, Los Angeles, California
  - Teva Investigational Site 5, Los Angeles, California
  - Teva Investigational Site 7, San Diego, California
  - Teva Investigational Site 14, San Leandro, California
  - Teva Investigational Site 17, Stanford, California
  - Teva Investigational Site 30, Aurora, Colorado
  - Teva Investigational Site 4, Aventura, Florida
  - Teva Investigational Site 32, Clearwater, Florida
  - Teva Investigational Site 35, Fort Lauderdale, Florida
  - Teva Investigational Site 1, Jupiter, Florida
  - Teva Investigational Site 11, Tampa, Florida
  - Teva Investigational Site 8, Atlanta, Georgia
  - Teva Investigational Site 31, Atlanta, Georgia
  - Teva Investigational Site 38, Stockbridge, Georgia
  - Teva Investigational Site 23, Coeur d'Alene, Idaho
  - Teva Investigational Site 37, Lexington, Kentucky
  - Teva Investigational Site 36, Baltimore, Maryland
  - Teva Investigational Site 10, Boston, Massachusetts
  - Teva Investigational Site 22, Ann Arbor, Michigan
  - Teva Investigational Site 9, Manhasset, New York
  - Teva Investigational Site 3, Chapel Hill, North Carolina
  - Teva Investigational Site 28, Charlotte, North Carolina
  - Teva Investigational Site 18, Durham, North Carolina
  - Teva Investigational Site 2, Monroe, North Carolina
  - Teva Investigational Site 21, Oklahoma City, Oklahoma
  - Teva Investigational Site 25, Duncansville, Pennsylvania
  - Teva Investigational Site 26, Pittsburgh, Pennsylvania
  - Teva Investigational Site 15, Charleston, South Carolina
  - Teva Investigational Site 29, Dallas, Texas
  - Teva Investigational Site 40, Houston, Texas
  - Teva Investigational Site 6, Houston, Texas
  - Teva Investigational Site 39, Mesquite, Texas
  - Teva Investigational Site 34, San Antonio, Texas
  - Teva Investigational Site 24, Temple, Texas
  - Teva Investigational Site 19, Arlington, Virginia
  - Teva Investigational Site 12, Seattle, Washington
  - Teva Investigational Site 33, Milwaukee, Wisconsin
- Belgium (3):
  - Teva Investigational Site 102, Brussels
  - Teva Investigational Site 101, Liège
  - Teva Investigational Site 100, Yvoir
- Czechia (4):
  - Teva Investigational Site 201, Brno
  - Teva Investigational Site 200, Olomouc
  - Teva Investigational Site 202, Prague
  - Teva Investigational Site 203, Prague
- France (5):
  - Teva Investigational Site 301, Lille
  - Teva Investigational Site 302, Nantes
  - Teva Investigational Site 300, Paris
  - Teva Investigational Site 303, Paris
  - Teva Investigational Site 304, Strasbourg
- Germany (7):
  - Teva Investigational Site 402, Aachen
  - Teva Investigational Site 403, Berlin
  - Teva Investigational Site 401, Dresden
  - Teva Investigational Site 404, Düsseldorf
  - Teva Investigational Site 406, Hamburg
  - Teva Investigational Site 405, Mainz
  - Teva Investigational Site 400, München
- Hungary (3):
  - Teva Investigational Site 501, Budapest
  - Teva Investigational Site 502, Debrecen
  - Teva Investigational Site 500, Zalaegerszeg
- Poland (7):
  - Teva Investigational Site 603, Dąbrówka
  - Teva Investigational Site 600, Elblag
  - Teva Investigational Site 602, Gmina Końskie
  - Teva Investigational Site 604, Lublin
  - Teva Investigational Site 601, Lublin
  - Teva Investigational Site 606, Warsaw
  - Teva Investigational Site 605, Wroclaw
- Portugal (4):
  - Teva Investigational Site 701, Amadora
  - Teva Investigational Site 702, Coimbra
  - Teva Investigational Site 703, Porto
  - Teva Investigational Site 700, Porto
- Spain (3):
  - Teva Investigational Site 751, Dresden
  - Teva Investigational Site 752, Santander
  - Teva Investigational Site 750, Seville
- Ukraine (6):
  - Teva Investigational Site 901, Donetsk
  - Teva Investigational Site 905, Ivano-Frankivsk
  - Teva Investigational Site 900, Kyiv
  - Teva Investigational Site 902, Kyiv
  - Teva Investigational Site 903, Kyiv
  - Teva Investigational Site 904, Lviv
- United Kingdom (4):
  - Teva Investigational Site 803, Bath
  - Teva Investigational Site 801, Leeds
  - Teva Investigational Site 800, London
  - Teva Investigational Site 802, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Groups:
- CEP-33457: Participants received 200 micrograms (mcg) of CEP-33457 subcutaneously (SC) every 4 weeks for a maximum of 17 doses (64 weeks).
Period: Overall Study
Arm/Group | CEP-33457
Started | 136
Received at Least 1 Dose of Study Drug | 136
Completed | 1
Not Completed | 135
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 2
Not completed — Other than specified | 3
Not completed — Withdrawn due to early study termination | 107

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set included all participants who were enrolled in the study, regardless of whether or not a participant took any study drug.
Groups:
- CEP-33457: Participants received 200 mcg of CEP-33457 SC every 4 weeks for a maximum of 17 doses (64 weeks).
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 101
  Race: Black | 22
  Race: Asian | 5
  Race: Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included clinically significant vitals, labs, and physical examination findings. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 72
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants | 117

2. Secondary Outcome: Number of Participants Achieving a Clinical Response Using the Systemic Lupus Erythematosus (SLE) Responder Index (SRI)
Description: An SRI response was defined as a reduction from baseline in SLE Disease Activity Index 2000 (SLEDAI-2K) score of ≥4 points, no worsening in Physician Global Assessment (PhGA), no new British Isles Lupus Assessment Group (BILAG) A body system score, and ≤1 new BILAG B body system score from baseline. SLEDAI 2K includes 24 weighted clinical and laboratory variables. Total score = 0 to 105. A score of 6 to 10 = moderate disease activity, and a reduction of >3 points = improvement. PhGA was completed by physician using a visual analog scale (VAS) from 0=none to 3=severe. A change of >0.3 points = worsening. BILAG includes 97 clinical and laboratory items. Each organ system is assigned a score displayed as a grade from A to E: A=very active disease; B=participant needs increase in treatment for moderately active disease; C=stable or mild disease; D=previous organ involvement but no current disease activity; and E=no current disease activity and organ system has never been involved.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: Intent-to-treat (ITT) analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  Week 4 | 10
  Week 8 | 18
  Week 12 | 19
  Week 16 | 19
  Week 20 | 21
  Week 24 | 18
  Week 28 | 17
  Week 32 | 11
  Week 36 | 12
  Week 40 | 10
  Week 44 | 6
  Week 48 | 5
  Week 52 | 5
  Week 56 | 6
  Week 60 | 2
  Week 64 | 1
  Week 68 | 0
  Week 72 | 0

3. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Total Score
Description: The SLEDAI-2K is a validated objective measure that assesses disease activity within the last 28 days before completion of the index. It is a global index and includes 24 weighted clinical and laboratory variables. The total score (sum of all 24 scores) ranges from 0 to 105, with higher scores representing increased disease activity.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64 and Final Assessment (or Early Termination [up to Week 72])
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
units on a scale
  Change at Week 4: number analyzed (Participants) | 127
  Change at Week 4 | -0.4 (2.48)
  Change at Week 8: number analyzed (Participants) | 122
  Change at Week 8 | -0.9 (2.36)
  Change at Week 12: number analyzed (Participants) | 118
  Change at Week 12 | -0.9 (2.71)
  Change at Week 16: number analyzed (Participants) | 113
  Change at Week 16 | -0.7 (2.74)
  Change at Week 20: number analyzed (Participants) | 91
  Change at Week 20 | -1.3 (3.10)
  Change at Week 24: number analyzed (Participants) | 59
  Change at Week 24 | -1.5 (3.40)
  Change at Week 28: number analyzed (Participants) | 47
  Change at Week 28 | -2.0 (3.80)
  Change at Week 32: number analyzed (Participants) | 36
  Change at Week 32 | -1.9 (3.48)
  Change at Week 36: number analyzed (Participants) | 32
  Change at Week 36 | -2.1 (3.39)
  Change at Week 40: number analyzed (Participants) | 29
  Change at Week 40 | -1.9 (3.34)
  Change at Week 44: number analyzed (Participants) | 25
  Change at Week 44 | -2.3 (3.84)
  Change at Week 48: number analyzed (Participants) | 21
  Change at Week 48 | -2.2 (3.86)
  Change at Week 52: number analyzed (Participants) | 17
  Change at Week 52 | -3.0 (3.94)
  Change at Week 56: number analyzed (Participants) | 13
  Change at Week 56 | -3.6 (4.41)
  Change at Week 60: number analyzed (Participants) | 8
  Change at Week 60 | -2.3 (5.52)
  Change at Week 64: number analyzed (Participants) | 4
  Change at Week 64 | -3.3 (6.50)
  Change at Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 134
  Change at Final Assessment (or Early Termination [up to Week 72]) | -0.9 (3.62)

4. Secondary Outcome: Number of Participants With British Isles Lupus Assessment Group 2004 (BILAG-2004) Response
Description: The BILAG-2004 is a validated objective and subjective global measure of the SLE disease activity, based on the physician's intention to treat, and refers to disease activity within the last 4 weeks before completion of the index. It includes 97 clinical and laboratory components to evaluate SLE disease activity in 9 different body systems (constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal, and hematological). Each body system is assigned a score displayed as a grade from A to E, as follows: A=very active disease; B=participant needs increase in treatment for moderately active disease; C=stab1e or mild disease; D=previous system involvement but no current disease activity; and E=no current disease activity and the body system has never been involved. BILAG 2004 response was defined as no new BILAG A body system score and no more than 1 new BILAG B body system score from baseline.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  Week 4 | 126
  Week 8 | 118
  Week 12 | 111
  Week 16 | 110
  Week 20 | 88
  Week 24 | 56
  Week 28 | 47
  Week 32 | 34
  Week 36 | 30
  Week 40 | 28
  Week 44 | 22
  Week 48 | 19
  Week 52 | 15
  Week 56 | 12
  Week 60 | 7
  Week 64 | 3
  Week 68 | 0
  Week 72 | 0

5. Secondary Outcome: Number of Participants Showing No Worsening on Physician's Global Assessment (PhGA) Scale
Description: The PhGA was completed by the physician using a 3-inch visual analog scale (VAS) labeled from 0=none to 3=severe. A change of greater than 0.3 point on the VAS indicates worsening. The number of participants showing no worsening are presented.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  Week 4 | 113
  Week 8 | 111
  Week 12 | 105
  Week 16 | 100
  Week 20 | 76
  Week 24 | 48
  Week 28 | 41
  Week 32 | 34
  Week 36 | 28
  Week 40 | 25
  Week 44 | 20
  Week 48 | 19
  Week 52 | 15
  Week 56 | 10
  Week 60 | 8
  Week 64 | 3
  Week 68 | 0
  Week 72 | 0

6. Secondary Outcome: Number of Participants Showing No Worsening on Patient's Global Assessment (PtGA) Scale
Description: The PtGA was completed by the participant, using a 3-inch VAS labeled from 0=none to 3=severe. A change of greater than 0.3 point on the VAS indicated worsening. The number of participants showing no worsening are presented.
Time Frame: Week 12, 24, 36, 48, 60, and 72
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  Week 12 | 90
  Week 24 | 43
  Week 36 | 23
  Week 48 | 17
  Week 60 | 6
  Week 72 | 0

7. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Domain Scores
Description: The SF-36 questionnaire has 36 questions composing the scale that represent 8 domains: 1) physical functioning, 2) physical role functioning, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) emotional role functioning, and 8) mental health. All domains are scored on a scale from 0 (worst) to 100 (best), with higher scores representing the best possible health state. Change from baseline scores in the following individual standardized domains: Bodily pain, physical functioning, social functioning and vitality were presented.
Time Frame: Baseline, Week 12, 24, 36, 48, 60 and final assessment (or early termination [up to Week 72])
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CEP-33457
Number analyzed (Participants) | 134
units on a scale
  Bodily pain: Change at Week 12: number analyzed (Participants) | 118
  Bodily pain: Change at Week 12 | 2.8 (16.43)
  Bodily pain: Change at Week 24: number analyzed (Participants) | 59
  Bodily pain: Change at Week 24 | 1.5 (20.68)
  Bodily pain: Change at Week 36: number analyzed (Participants) | 32
  Bodily pain: Change at Week 36 | 5.5 (23.09)
  Bodily pain: Change at Week 48: number analyzed (Participants) | 20
  Bodily pain: Change at Week 48 | 8.8 (16.18)
  Bodily pain: Change at Week 60: number analyzed (Participants) | 8
  Bodily pain: Change at Week 60 | 9.0 (28.59)
  Bodily pain: Change at Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 133
  Bodily pain: Change at Final Assessment (or Early Termination [up to Week 72]) | 2.7 (20.26)
  Physical functioning: Change at Week 12: number analyzed (Participants) | 118
  Physical functioning: Change at Week 12 | 1.7 (12.28)
  Physical functioning: Change at Week 24: number analyzed (Participants) | 59
  Physical functioning: Change at Week 24 | -0.4 (15.57)
  Physical functioning: Change at Week 36: number analyzed (Participants) | 32
  Physical functioning: Change at Week 36 | -0.5 (17.20)
  Physical functioning: Change at Week 48: number analyzed (Participants) | 20
  Physical functioning: Change at Week 48 | 3.0 (14.36)
  Physical functioning: Change at Week 60: number analyzed (Participants) | 8
  Physical functioning: Change at Week 60 | 4.4 (15.45)
  Physical functioning: Change at Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 133
  Physical functioning: Change at Final Assessment (or Early Termination [up to Week 72]) | 1.1 (17.04)
  Social functioning: Change at Week 12: number analyzed (Participants) | 118
  Social functioning: Change at Week 12 | 0.7 (15.18)
  Social functioning: Change at Week 24: number analyzed (Participants) | 59
  Social functioning: Change at Week 24 | 3.6 (19.43)
  Social functioning: Change at Week 36: number analyzed (Participants) | 32
  Social functioning: Change at Week 36 | 2.3 (21.87)
  Social functioning: Change at Week 48: number analyzed (Participants) | 20
  Social functioning: Change at Week 48 | -0.6 (22.75)
  Social functioning: Change at Week 60: number analyzed (Participants) | 8
  Social functioning: Change at Week 60 | 7.8 (21.06)
  Social functioning: Change at Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 133
  Social functioning: Change at Final Assessment (or Early Termination [up to Week 72]) | -0.1 (20.56)
  Vitality: Change at Week 12: number analyzed (Participants) | 118
  Vitality: Change at Week 12 | 3.4 (15.28)
  Vitality: Change at Week 24: number analyzed (Participants) | 59
  Vitality: Change at Week 24 | 2.1 (18.04)
  Vitality: Change at Week 36: number analyzed (Participants) | 32
  Vitality: Change at Week 36 | 3.9 (19.03)
  Vitality: Change at Week 48: number analyzed (Participants) | 20
  Vitality: Change at Week 48 | 4.7 (17.78)
  Vitality: Change at Week 60: number analyzed (Participants) | 8
  Vitality: Change at Week 60 | 7.0 (23.25)
  Vitality: Change at Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 133
  Vitality: Change at Final Assessment (or Early Termination [up to Week 72]) | 2.6 (15.94)

8. Secondary Outcome: Change From Baseline in the Biomarker: Anti-U1 Ribonucleoprotein Antibody (Anti-UI RNP Ab)
Description: Anti-UI RNP Ab was measured from blood serum collected at specified time points.
Time Frame: Baseline, Week 12, 24, 36, 48, 60 and final assessment (or early termination [up to Week 72])
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'number analyzed' signifies participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units (U)/milliliter (mL)
Arm/Group | CEP-33457
Number analyzed (Participants) | 132
units (U)/milliliter (mL)
  Change at Week 12: number analyzed (Participants) | 115
  Change at Week 12 | 193.0 (505.20)
  Change at Week 24: number analyzed (Participants) | 58
  Change at Week 24 | 313.6 (642.69)
  Change at Week 36: number analyzed (Participants) | 30
  Change at Week 36 | 199.2 (497.79)
  Change at Week 48: number analyzed (Participants) | 21
  Change at Week 48 | 327.7 (643.54)
  Change at Week 60: number analyzed (Participants) | 8
  Change at Week 60 | 480.1 (723.53)
  Change at Final Assessment (or Early Termination [up to Week 72]) | 154.7 (470.23)

9. Secondary Outcome: Change From Baseline in the Biomarker: C-Reactive Protein (CRP)
Description: CRP was measured from blood serum samples at specified time points.
Time Frame: Baseline, Week 12, 24, 36, 48, 60, and Final Assessment (or Early Termination [up to Week 72])
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams (mg)/deciliter (dL)
Arm/Group | CEP-33457
Number analyzed (Participants) | 132
milligrams (mg)/deciliter (dL)
  Change at Week 12: number analyzed (Participants) | 117
  Change at Week 12 | 0 (0.68)
  Change at Week 24: number analyzed (Participants) | 59
  Change at Week 24 | 0 (0.48)
  Change at Week 36: number analyzed (Participants) | 30
  Change at Week 36 | -0.1 (0.41)
  Change at Week 48: number analyzed (Participants) | 21
  Change at Week 48 | 0 (0.46)
  Change at Week 60: number analyzed (Participants) | 8
  Change at Week 60 | -0.1 (0.30)
  Change at Final Assessment (or Early Termination [up to Week 72]) | 0 (0.82)

10. Secondary Outcome: Number of Participants With Anti-nuclear Antibodies (ANA)
Description: Anti-nuclear antibodies (ANA) were measured from blood serum samples at specified time points.
Time Frame: Week 12, 24, 36, 48, 60, and Final Assessment (or Early Termination [up to Week 72])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 126
Participants
  Week 12: number analyzed (Participants) | 112
  Week 12: None detected | 0
  Week 12: <1:40 | 0
  Week 12: 1:40 | 16
  Week 12: 1:80 | 17
  Week 12: 1:160 | 20
  Week 12: 1:320 | 30
  Week 12: 1:640 | 7
  Week 12: 1:1280 | 0
  Week 12: >=1:1280 | 22
  Week 24: number analyzed (Participants) | 57
  Week 24: None detected | 0
  Week 24: <1:40 | 0
  Week 24: 1:40 | 3
  Week 24: 1:80 | 11
  Week 24: 1:160 | 12
  Week 24: 1:320 | 11
  Week 24: 1:640 | 4
  Week 24: 1:1280 | 0
  Week 24: >=1:1280 | 16
  Week 36: number analyzed (Participants) | 30
  Week 36: None detected | 0
  Week 36: <1:40 | 0
  Week 36: 1:40 | 5
  Week 36: 1:80 | 6
  Week 36: 1:160 | 7
  Week 36: 1:320 | 4
  Week 36: 1:640 | 2
  Week 36: 1:1280 | 0
  Week 36: >=1:1280 | 6
  Week 48: number analyzed (Participants) | 20
  Week 48: None detected | 0
  Week 48: <1:40 | 0
  Week 48: 1:40 | 4
  Week 48: 1:80 | 4
  Week 48: 1:160 | 3
  Week 48: 1:320 | 2
  Week 48: 1:640 | 2
  Week 48: 1:1280 | 0
  Week 48: >=1:1280 | 5
  Week 60: number analyzed (Participants) | 8
  Week 60: None detected | 0
  Week 60: <1:40 | 0
  Week 60: 1:40 | 1
  Week 60: 1:80 | 2
  Week 60: 1:160 | 2
  Week 60: 1:320 | 1
  Week 60: 1:640 | 1
  Week 60: 1:1280 | 0
  Week 60: >=1:1280 | 1
  Final Assessment (or Early Termination [up to Week 72]): None detected | 0
  Final Assessment (or Early Termination [up to Week 72]): <1:40 | 0
  Final Assessment (or Early Termination [up to Week 72]): 1:40 | 16
  Final Assessment (or Early Termination [up to Week 72]): 1:80 | 16
  Final Assessment (or Early Termination [up to Week 72]): 1:160 | 18
  Final Assessment (or Early Termination [up to Week 72]): 1:320 | 28
  Final Assessment (or Early Termination [up to Week 72]): 1:640 | 18
  Final Assessment (or Early Termination [up to Week 72]): 1:1280 | 0
  Final Assessment (or Early Termination [up to Week 72]): >=1:1280 | 30

11. Secondary Outcome: Number of Participants With Mild to Moderate Flare, Severe Flare, and No Flare, Based on the Safety of Estrogens in Lupus Erythematosus: National Assessment (SELENA) Flare Index
Description: The SELENA Flare Index divides flares into 2 categories: mild/moderate and severe. A severe flare would lead to early withdrawal. The number of participants with mild to moderate flare, severe flare, and no flare at each visit during the treatment period were reported.
Time Frame: Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64 and Final Assessment (or Early Termination [up to Week 72])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 135
Participants
  Week 4: number analyzed (Participants) | 130
  Week 4: Mild/moderate flare | 15
  Week 4: Severe flare | 1
  Week 4: No flare | 114
  Week 8: number analyzed (Participants) | 122
  Week 8: Mild/moderate flare | 13
  Week 8: Severe flare | 0
  Week 8: No flare | 109
  Week 12: number analyzed (Participants) | 118
  Week 12: Mild/moderate flare | 21
  Week 12: Severe flare | 0
  Week 12: No flare | 97
  Week 16: number analyzed (Participants) | 113
  Week 16: Mild/moderate flare | 14
  Week 16: Severe flare | 0
  Week 16: No flare | 99
  Week 20: number analyzed (Participants) | 91
  Week 20: Mild/moderate flare | 9
  Week 20: Severe flare | 0
  Week 20: No flare | 82
  Week 24: number analyzed (Participants) | 59
  Week 24: Mild/moderate flare | 8
  Week 24: Severe flare | 0
  Week 24: No flare | 51
  Week 28: number analyzed (Participants) | 47
  Week 28: Mild/moderate flare | 8
  Week 28: Severe flare | 0
  Week 28: No flare | 39
  Week 32: number analyzed (Participants) | 37
  Week 32: Mild/moderate flare | 5
  Week 32: Severe flare | 0
  Week 32: No flare | 32
  Week 36: number analyzed (Participants) | 32
  Week 36: Mild/moderate flare | 4
  Week 36: Severe flare | 0
  Week 36: No flare | 28
  Week 40: number analyzed (Participants) | 29
  Week 40: Mild/moderate flare | 4
  Week 40: Severe flare | 0
  Week 40: No flare | 25
  Week 44: number analyzed (Participants) | 25
  Week 44: Mild/moderate flare | 4
  Week 44: Severe flare | 0
  Week 44: No flare | 21
  Week 48: number analyzed (Participants) | 21
  Week 48: Mild/moderate flare | 2
  Week 48: Severe flare | 0
  Week 48: No flare | 19
  Week 52: number analyzed (Participants) | 17
  Week 52: Mild/moderate flare | 2
  Week 52: Severe flare | 0
  Week 52: No flare | 15
  Week 56: number analyzed (Participants) | 13
  Week 56: Mild/moderate flare | 3
  Week 56: Severe flare | 0
  Week 56: No flare | 10
  Week 60: number analyzed (Participants) | 8
  Week 60: Mild/moderate flare | 2
  Week 60: Severe flare | 0
  Week 60: No flare | 6
  Week 64: number analyzed (Participants) | 4
  Week 64: Mild/moderate flare | 1
  Week 64: Severe flare | 0
  Week 64: No flare | 3
  Final Assessment (or Early Termination [up to Week 72]): Mild/moderate flare | 24
  Final Assessment (or Early Termination [up to Week 72]): Severe flare | 4
  Final Assessment (or Early Termination [up to Week 72]): No flare | 107

12. Secondary Outcome: Change From Baseline in Total Damage Score as Assessed by the Systemic Lupus International Collaborative Clinics/American College of Rheumatology (SLICC/ACR) Damage Index
Description: The SLICC/ACR damage index assesses specific comorbidities associated with SLE. It consists of 41 items and covers 12 body systems. Total damage scores were calculated using the 41 items. The total damage score ranges from 0 (no damage) to 47 (maximum disease damage severity) with higher scores indicating increasing disease damage severity.
Time Frame: Baseline, Week 24, 48 and Final Assessment (or Early Termination [up to Week 72])
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CEP-33457
Number analyzed (Participants) | 133
units on a scale
  Change at Week 24: number analyzed (Participants) | 59
  Change at Week 24 | 0 (0.42)
  Change at Week 48: number analyzed (Participants) | 21
  Change at Week 48 | -0.1 (0.48)
  Change at Final Assessment (or Early Termination [up to Week 72]) | -0.1 (0.44)

13. Secondary Outcome: Number of Participants Achieving Remission of Disease
Description: Remission of disease was defined as a reduction of SLEDAI-2K score to 0. The SLEDAI-2K is a validated objective measure that assesses disease activity within the last 28 days before completion of the index. It is a global index and includes 24 weighted clinical and laboratory variables. The total score (sum of all 24 scores) ranges from 0 to 105, with higher scores representing increased disease activity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64 and Final Assessment (or Early Termination [up to Week 72])
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug. Here 'number analyzed' signifies participants evaluable at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  Week 4: number analyzed (Participants) | 130
  Week 4 | 8
  Week 8: number analyzed (Participants) | 122
  Week 8 | 9
  Week 12: number analyzed (Participants) | 118
  Week 12 | 11
  Week 16: number analyzed (Participants) | 113
  Week 16 | 10
  Week 20: number analyzed (Participants) | 91
  Week 20 | 10
  Week 24: number analyzed (Participants) | 59
  Week 24 | 4
  Week 28: number analyzed (Participants) | 47
  Week 28 | 2
  Week 32: number analyzed (Participants) | 37
  Week 32 | 1
  Week 36: number analyzed (Participants) | 32
  Week 36 | 1
  Week 40: number analyzed (Participants) | 29
  Week 40 | 1
  Week 44: number analyzed (Participants) | 25
  Week 44 | 1
  Week 48: number analyzed (Participants) | 21
  Week 48 | 1
  Week 52: number analyzed (Participants) | 17
  Week 52 | 1
  Week 56: number analyzed (Participants) | 13
  Week 56 | 1
  Week 60: number analyzed (Participants) | 8
  Week 60 | 0
  Week 64: number analyzed (Participants) | 4
  Week 64 | 0
  Final Assessment (or Early Termination [up to Week 72]): number analyzed (Participants) | 134
  Final Assessment (or Early Termination [up to Week 72]) | 8

14. Secondary Outcome: Number of Participants With Change in Steroid Dose
Description: Number of participants with change in steroid dose (prednisone equivalent/day) were reported. The change in steroid dose was evaluated to determine the number of participants taking a dose less than 7.5 mg of prednisone equivalent/day, a dose of 7.5 mg prednisone equivalent/day or more, and none per day.
Time Frame: From Baseline up to Final Assessment (or Early Termination [up to Week 72])
Population: ITT analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants
  <7.5 mg at Baseline to <7.5 mg at Final Assessment | 37
  <7.5 mg at Baseline to >=7.5 mg at Final Assessment | 1
  <7.5 mg at Baseline to None at Final Assessment | 0
  >=7.5 mg at Baseline to <7.5 mg at Final Assessment | 5
  >=7.5 mg at Baseline to >=7.5 mg at Final Assessment | 49
  >=7.5 mg at Baseline to None at Final Assessment | 3
  None at Baseline to <7.5 mg at Final Assessment | 3
  None at Baseline to >=7.5 mg at Final Assessment | 2
  None at Baseline to None at Final Assessment | 36

15. Secondary Outcome: Number of Participants With Reactive and Non-Reactive Anti-CEP-33457 Antibodies
Description: Immunogenicity was assessed by detection of the presence of specific anti-CEP-33457 antibodies in blood serum samples collected at the specified time points.
Time Frame: Week 24, 48 and Final Assessment (or Early Termination [up to Week 72])
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 126
Participants
  Week 24: number analyzed (Participants) | 57
  Week 24: Reactive | 4
  Week 24: Non-reactive | 53
  Week 48: number analyzed (Participants) | 22
  Week 48: Reactive | 1
  Week 48: Non-reactive | 21
  Final Assessment (or Early Termination [up to Week 72]): Reactive | 7
  Final Assessment (or Early Termination [up to Week 72]): Non-reactive | 119

16. Primary Outcome: Number of Participants Who Received Concomitant Medications
Description: Any concomitant therapy or medication taken while the participant received study drug.
Time Frame: Baseline up to Week 72
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CEP-33457
Number analyzed (Participants) | 136
Participants | 136

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: Safety analysis set included all enrolled participants who took at least 1 dose of study drug.
Arm/Group | CEP-33457
All-Cause Mortality (participants affected / at risk) | 0/136
Serious Adverse Events (participants affected / at risk) | 11/136
Other Adverse Events (participants affected / at risk) | 89/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-33457 (N=136)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEP-33457 (N=136)
Diarrhoea (Gastrointestinal disorders) | 10 (17)
Nausea (Gastrointestinal disorders) | 10 (12)
Bronchitis (Infections and infestations) | 8 (9)
Nasopharyngitis (Infections and infestations) | 11 (13)
Sinusitis (Infections and infestations) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 20 (25)
Urinary tract infection (Infections and infestations) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 15 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 18 (26)
Headache (Nervous system disorders) | 10 (16)
Anxiety (Psychiatric disorders) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 16 (17)

LIMITATIONS AND CAVEATS:
The study was terminated early due to business decision; there were no safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.